CLINICAL TRIAL: NCT01934972
Title: A Randomized Controlled Trial of Cognitive Remediation and D-cycloserine for Individuals With Bipolar Disorder
Acronym: DCS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Nicholas Breitborde, Assistant Professor, Psychiatry, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-0926-01 Breitborde DCS
Record Dates: First submitted 2013-08-19; First posted 2013-09-04 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Cycloserine; Cognitive Remediation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CR + DCS (Experimental): Subjects will receive Cognitive Remediation and active study drug.
  Interventions: Other: CR + DCS (D-cycloserine)
- CR + placebo (Active Comparator): Cognitive Remediation and placebo
  Interventions: Other: CR + placebo

INTERVENTIONS:
Other: CR + DCS (D-cycloserine) — CR + DCS
  Other Names: DCS and Cognitive Remediation
  Arms: CR + DCS
Other: CR + placebo — CR + placebo
  Other Names: Cognitive Remediation
  Arms: CR + placebo

SUMMARY:
Individuals with bipolar suffer from problems in basic cognitive skills such as memory and concentration. Unfortunately, there are no current treatments that have been shown to improve cognitive skills among individuals with bipolar disorder.

Computerized cognitive remediation (CR) is a treatment that has been shown to improve cognitive skills among individuals with serious mental illnesses other than bipolar disorder, such as schizophrenia. This treatment involves completing a series of activities on a computer that have been shown to improve cognitive skills.

D-cycloserine (DCS) is an antibiotic traditionally used in the treatment of tuberculosis. Recent studies have suggested that this drug may also improve individuals' ability to learn. Thus, the goal of our study is to examine whether receipt of d-cycloserine increases the benefit that individuals receive from participation in cognitive remediation.

To test this hypothesis, approximately forty subjects will be randomized to one of two study arms: [i] CR + DCS or [ii] CR + placebo. We will examine whether d-cycloserine increases the benefit that individuals with bipolar disorder receive from participation in cognitive remediation.

DETAILED DESCRIPTION:
Individuals with bipolar disorder suffer from a broad array of cognitive deficits that may hinder their ability to achieve successful community functioning. Consequently, greater attention has recently been directed toward the development of strategies to ameliorate these cognitive deficits. One strategy which has been shown to be successful in this endeavor is cognitive remediation (CR). This intervention, which is recognized as a "best practice" in the treatment of serious mental illness, is typically comprised of a series of repeated exercises delivered by a clinician or via a computer that are designed to improve performance in cognitive functioning. Yet, despite the promise of cognitive remediation, the benefit of this intervention among individuals with bipolar disorder has yet to be investigated.

Recently, studies have demonstrated that d-cycloserine (DCS), an N-methyl-D-aspartate receptor (NMDAR) agonist, may facilitate the learning process for emotional and non-emotional information in both humans and animals. These results raise the possibility that DCS may increase the benefits associated with the receipt of cognitive remediation among individuals with bipolar disorder. To date, we are unaware of any study which has examined whether concurrent receipt of DCS may increase the benefits produced by cognitive remediation among individuals with a severe mental illness.

Thus, we propose to complete an exploratory investigation of augmenting cognitive remediation with DCS among individuals with bipolar disorder. Approximately forty subjects will be randomized to one of two study arms: [i] CR + DCS; or [ii] CR + placebo. The primary outcome of interest will be changes in cognitive functioning before and after receipt of the cognitive remediation intervention. Secondary outcomes of interest will be changes in symptomatology, social and vocational functioning, and performance of tasks of everyday living.

ELIGIBILITY:
- Inclusion Criteria: [i] Diagnosis of Bipolar I or Bipolar II Disorder determined by the Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders (DSM) [ii] Ages 18-65 [iii] No evidence of mental retardation, dementia, or other organic disorder that may reduce cognitive functioning [iv] premorbid intelligence quotient (IQ) greater than or equal to 70 as determined by reading subtest of the Wide Range Achievement Test.

[v] Able to provide informed consent as evidenced by passing the informed consent quiz with a score of 80% or greater.

[vi] Fluent in English as assessed per self-report from participant [vii] Female subjects cannot be pregnant or breastfeeding. All subjects must consent to using at least one form of birth control during study participation.

[viii] Current remission of depressive symptoms as indicated by a score of 8 or less on the Bipolar Depression Rating Scale.

[ix] Current remission of manic symptoms as indicated by a score of 7 or less on the Young Mania Scale

Exclusion criteria:

[i] Hypersensitivity to previous receipt of cycloserine per subject report [ii] Epilespy or history of seizures as assessed using the Medical History form [iii] Meets DSM-IV criteria for alcohol or drug abuse in the past month or dependence in the past three months.

[iv] Active suicidal or homicidal ideation [v] Initiation or increase in dosage of any antidepressant within six weeks, or mood stabilizer within four weeks as assessed using the Medication Checklist.

[vi] Previous or current participation in cognitive remediation per subject report [vii] Currently taking d-cycloserine [viii] Reduced kidney or liver functioning, vitamin B12 deficiency, folic acid deficiency, megaloblastic anemia, or sideroblastic anemia per baseline safety labs.

[ix] Currently taking medication known to have problematic interactions with d-cycloserine, including etionamide and isoniazid.

[x] History of the blood disease porphyria as assessed using the Medical History form [xi] Current active symptoms of psychosis defined as not meeting existing guidelines [12] for remission of psychotic symptoms using the Positive and Negative Syndrome Scale.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Breitborde, PhD, Principal Investigator — The University of Arizona
Locations (1):
- University of Arizona Medical Center South Campus, Tucson, Arizona, United States

REFERENCES:
- [Derived] Breitborde NJ, Dawson SC, Woolverton C, Dawley D, Bell EK, Norman K, Polsinelli A, Bernstein B, Mirsky P, Pletkova C, Grucci F 3rd, Montoya C, Nanadiego B, Sarabi E, DePalma M, Moreno F. A randomized controlled trial of cognitive remediation and d-cycloserine for individuals with bipolar disorder. BMC Psychol. 2014 Oct 10;2(1):41. doi: 10.1186/s40359-014-0041-4. eCollection 2014. PMID 25566387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment ended early due to the PI leaving the institution where the research was being completed (i.e., University of Arizona). Thus, only 23 people were enrolled in the study.
Pre-assignment Details: Six individuals of the 30 who were screened were not assigned to either of the intervention conditions. Four of these individuals dropped out prior to randomization to study arm. One was excluded due to an uncontrolled eating disorder, and one was excluded due to kidney dysfunction.
Period: Overall Study
Arm/Group | CR + DCS | CR + Placebo
Started | 13 | 11
Completed | 4 | 5
Not Completed | 9 | 6
Not completed — Withdrawal by Subject | 9 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CR + DCS | CR + Placebo | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.54 (15.83) | 41.1186 (15.22) | 42.97 (15.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 13 | 11 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 13 | 11 | 24
Region of Enrollment [Number; unit: participants]
  United States | 13 | 11 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Cognitive Functioning
Description: Level of cognitive functioning will be assessed via overall cognitive composite score from the Measurement and Treatment Research to Improve Cognition in Schizophrenia (MATRICS) Consensus Cognitive Battery. Scores on the MATRICS are presented at T-scores with a mean of 50 and standard deviation of 10 as compared to a normative sample. The possible range of scores are 0-100. Higher scores are indicative of better cognitive functioning.
  Change from baseline in cognitive functioning was calculated by taking the MATRICS overall cognitive functioning score at 26-week follow-up and subtracting the MATRICS overall cognitive composite score from baseline. Positive values on this score are indicative of improvements in cognitive functioning from baseline.
  Missing values on the MATRICS were addressed using multiple imputation
Time Frame: 26 weeks
Population: Missing data for this variable were addressed using multiple imputation. As such, the sample size for this measure is larger than for other measures listed below.
Measure: Mean (Standard Deviation); unit: T-Scores
Arm/Group | CR + DCS | CR + Placebo
Number analyzed (Participants) | 12 | 11
T-Scores | 10.90 (22.02) | 7.12 (8.72)

2. Secondary Outcome: Change From Baseline in Manic Symptomatology
Description: Manic symptomatology assesed using the Yung Mania Scale. Total scores on this scale range from 0 to 60 with higher scores indicative of greater severity of manic symptoms. Change scores from baseline were calculated by subtracting baseline total scores on this measure from 26-week scores. For this change score, positive values indicate that manic symptom severity was worse at 26-week follow-up than at baseline
Time Frame: 26 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR + DCS | CR + Placebo
Number analyzed (Participants) | 12 | 11
units on a scale | 0.27 (31.39) | -0.25 (6.60)

3. Secondary Outcome: Change From Baseline in Depressive Symptomatology
Description: Depressive symptomatology assessed using the Inventory of Depressive Symptomatology (Clinician-Rated). Total scores on this measure range from 0-84 with higher scores indicative of worse depressive symptomatology. Change from baseline in depressive symptomatology was calculated by subtracting baseline scores on the Inventory of Depressive Symptomatology from 26-week scores on this measure. Positive values of this change score indicate that depressive symptoms were worse at 26-week assessment than at baseline assessment.
Time Frame: 26 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR + DCS | CR + Placebo
Number analyzed (Participants) | 4 | 3
units on a scale | 1.25 (1.26) | 2.67 (8.08)

4. Secondary Outcome: Change From Baseline in Social Functioning
Description: Social functioning assessed using the Social Functioning Scale. Total score calculated by converting all subscale scores to a standard score with mean = 100 and standard deviation = 15. These subscale scores are then averaged to calculate the total score. There is no set minimum or maximum on this scale given this scoring procedure.
  Change from baseline in social functioning was calculated by subtracting total scores at baseline assessment from total scores at 26-week. A positive value on this change score are indicative of better social functioning at 26-week assessment than at baseline.
Time Frame: 26 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CR + DCS | CR + Placebo
Number analyzed (Participants) | 4 | 4
score on a scale | 17.87 (51.63) | 30.85 (52.78)

5. Secondary Outcome: Change From Baseline in Functional Capacity
Description: Functional capacity assessed using the Brief University of California, San Diego Performance-Based Skills Assessment (UPSA). Scores range from 0-100 with higher scores indicative of greater functional capacity.
  Change score were calculated by subtracting baseline scores on the UPSA from scores from the 6-month assessment. Positive values are indicative of higher functional capacity at 26-week follow-up as compared to baseline assessment.
Time Frame: 26 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CR + DCS | CR + Placebo
Number analyzed (Participants) | 3 | 3
score on a scale | 9.59 (11.42) | -9.26 (24.79)

6. Other Pre Specified Outcome: Change From Baseline in Health-related Quality of Life
Description: Health-related quality of life assessed using the RAND 36-Item Health Survey. Data are converted to Quality Adjusted Life Years (QALY) which has a minimum of 0 and a maximum of 1. Higher scores are indicative of greater health-related quality of life.
  Change scores are calculated by subtracting baseline scores from scores from 26-week assessment. Positive values on this change score indicate that health-related quality of life was higher at 26-weeks than baseline.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR + DCS | CR + Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | 0.01 (0.06) | 0.11 (0.10)

7. Other Pre Specified Outcome: Change From Baseline in Medication Adherence
Description: Medication adherence assessed using the Medication Adherence Rating Scale. Higher scores on this measure are indicative of worse medication adherence. Scores on this scale range from 0-10.
  Change scores were calculated by subtracted scores on this measure at baseline from scores at 26-week assessment. Positive values on this change score are indicative of worse medication adherence at 26-week follow-up as opposed to baseline assessment.
Time Frame: 26 Weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CR + DCS | CR + Placebo
Number analyzed (Participants) | 3 | 4
score on a scale | 0 (1) | 0.5 (0.58)

8. Other Pre Specified Outcome: Change From Baseline in Quality of Life
Description: Quality of life assessed using the World Health Organization Quality of Life Scale. A total score was calculated by averaging scores for the four subscales on this measure. Range for this total score is 0-100 with higher scores indicative of greater quality of life.
  Change scores were calculated by subtracting baseline scores on this measure from week-26 scores. Positive values for this change score indicate the quality of life scores were greater at week 26 than at baseline.
Time Frame: 26 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CR + DCS | CR + Placebo
Number analyzed (Participants) | 3 | 3
units on a scale | 7.75 (8.23) | 7.92 (4.06)

9. Other Pre Specified Outcome: Change From Baseline in Stage of Recovery
Description: Stage of recovery assessed using the Stages of Recovery Instrument. This instrument identifies which phase of recovery the participant identifies themselves to be within: moratorium, awareness, preparation, rebuilding, and growth. Outcome presented in the number of participants identifying as being within the growth phase of recovery at 26-week followup
Time Frame: 26 weeks
Measure: Number; unit: participants
Arm/Group | CR + DCS | CR + Placebo
Number analyzed (Participants) | 3 | 3
participants | 2 | 2

10. Other Pre Specified Outcome: Change From Baseline in Metacognition
Description: Metacognition assessed using the Metacognitive Awareness Inventory. Total scores on this measure range from 0-100 with higher scores indicative of greater metacognition.
  Change in metacognition from baseline was calculated by subtracting baseline total scores on this measure from total scores on this measure at 26-week assessment. Positive values on this change score indicate that metacognition scores were higher at 26-week assessment than at baseline assessment
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CR + DCS | CR + Placebo
Number analyzed (Participants) | 2 | 2
score on a scale | 59.56 (48.22) | 57.04 (5.88)

11. Other Pre Specified Outcome: Change in Instrinsic Motivation From Baseline
Description: Intrinsic motivation assessed using the Intrinsic Motivation Inventory (IMI). Scores on this measure range from 21-147 with higher scores indicative of greater intrinsic motivation. For the current study, we asked specifically about intrinsic motivation to participate in CR.
  Change scores were calculated by subtracting baseline total scores on this measure from total scores obtained at 26-week assessment. Positive values on this change score indicate that participants reported greater intrinsic motivation as 26-week assessment as compared to baseline assessment.
Time Frame: 26 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CR + DCS | CR + Placebo
Number analyzed (Participants) | 2 | 3
score on a scale | 14.5 (12.02) | 7.67 (4.04)

12. Other Pre Specified Outcome: Frequency of Side Effects During Study Participation
Description: Assessed using the Systematic Assessment for Treatment Emergent Events. Number of participants who endorsed an adverse event during study participation
Time Frame: 26 Weeks
Measure: Number; unit: participants
Arm/Group | CR + DCS | CR + Placebo
Number analyzed (Participants) | 12 | 11
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant throughout the 6-month study duration
Arm/Group | CR + DCS | CR + Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/11
Other Adverse Events (participants affected / at risk) | 0/13 | 0/11

LIMITATIONS AND CAVEATS:
Study was terminated early due to PI leaving previous institution. A high number of participants did not complete full duration of study interventions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-10-10): https://cdn.clinicaltrials.gov/large-docs/72/NCT01934972/Prot_SAP_000.pdf